CLINICAL TRIAL: NCT04178759
Title: Impact of Chemotherapy and Regenerative Markers on Liver Regeneration After Liver Resection for Liver Metastases
Brief Title: Impact of Chemotherapy and Regenerative Markers of Liver Regeneration After Liver Resection for Liver Metastases
Acronym: VULSK-Hep
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vilnius University (Other)
Responsible Party: Principal Investigator, Kestutis Strupas, Chair of Department of Surgery, Vilnius University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019/3-1112-605
Record Dates: First submitted 2019-11-22; First posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Liver Regeneration; Liver Metastases
Keywords: Liver metastases; Liver regeneration; Markers
MeSH Terms: interventions — Hepatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Patients with benign liver disease, who undergo liver resection
  Interventions: Procedure: Liver resection
- Experimental (Experimental): Patients with liver metastases and received chemotherapy, who undergo liver resection
  Interventions: Procedure: Liver resection

INTERVENTIONS:
Procedure: Liver resection — Laparoscopic or open approach liver resection where at least 1 segment is removed

SUMMARY:
Liver is special organ, which can regenerate. On that ability there are many treatment modalities, where liver resection is performed, especially in cancer patients with liver metastases. Liver regeneration provides an opportunity for these patients to undergo multiple treatment regimes and liver resections to achieve curability. There are many factors that impair liver regeneration. One of these factors is chemotherapy. Literature data on impact of chemotherapy to liver regeneration is ambiguous. Therefore we aim to research impact of chemotherapy to liver regeneration.

DETAILED DESCRIPTION:
Liver is the largest parenchymal organ responsible for over 500 different functions in human body, which are detoxification of various toxins, drugs, synthesis of proteins and enzymes, coagulation factors. Liver is special organ, which can regenerate. If 75% of liver is removed it can regenerate to its normal size. Liver volume is very important to liver function, if there is volume insufficiency it could lead to liver failure in addition to other factors that impair liver regeneration. On that regenerative ability there are many treatment modalities, when liver resection is performed, especially in cancer patients with liver metastases. Modern treatment modalities are based on combination of different treatments, surgical and chemotherapeutic. On the other hand, side effects of chemotherapy should not be discarded, which can increase patient morbidity and mortality. Thus, liver regeneration provides an opportunity for these patients to undergo multiple treatment regimes and liver resections to achieve curability. Literature data on impact of chemotherapy to liver regeneration is ambiguous. Therefore we aim to research impact of chemotherapy to liver regeneration.

ELIGIBILITY:
Inclusion Criteria:

• Patients with liver lesions, who are eligible for liver resection

Exclusion Criteria:

* Pregnant women
* Liver resection is not performed

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Volume of regenerated liver after liver resection | 30 days
  Difference of liver volume preoperatively and postoperatively, meassured by CT

SECONDARY OUTCOMES:
Evaluation of liver fibrosis | 30 days
  The dynamic of liver fibrosis will be measured by ultrasound elastography pre-op and post-op day 1, 7 and 30;
Evaluation of liver markers responsible for liver regeneration | 30 days
  Expression of liver regeneration markers - hepatocyte growth factor and tumor growth factor beta1 - will be measured before and post-op day 1,3 and 7 in serum and also in liver tissue with immunohistochemistry
Evaluation of short term surgical outcomes | 90 days
  Complication rate will be assessed after 30 and 90 days post operatively

CONTACTS AND LOCATIONS:
Locations (1):
- Vilnius University Hospital Santaros Clinics, Vilnius, Lithuania